CLINICAL TRIAL: NCT02486510
Title: Effect of Cytoreductive Chemotherapy and a CCR5 Coreceptor Antagonist on HIV-1 Eradication
Acronym: CHEMOMAR
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Futility criteria
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHEMOMAR
Record Dates: First submitted 2015-06-24; First posted 2015-07-01 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: HIV-1 Infection
Keywords: HIV-1; CCR5 coreceptors; Maraviroc
MeSH Terms: interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Control) (No Intervention): Patients receiving intensive chemotherapy with/without stable antiretroviral therapy. Patients not receiving antiretroviral therapy will start it.
  Patients randomized to this group will not receive clinical trial treatment (neither Maraviroc or Placebo)
- Group 2 (Treatment) (Experimental): Patients receiving intensive chemotherapy with/without stable antiretroviral therapy and Maraviroc.
  Patients not receiving antiretroviral therapy will start this theraphy together with Maraviroc.
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — Patients randomized to experimental control will start Maraviroc treatment before, during and after chemotherapy until lymphocytes level recovery.
  Maraviroc Dose: 300 mg/12 hours For patients receiving an HIV-protease inhibitor (except tipranavir or Fosamprenavir), the dose will be reduced to 150 mg/12hours For patients receiving Efavirenz dose the dose will be 600 mg/12hours
  Other Names: Celsentri
  Arms: Group 2 (Treatment)

SUMMARY:
Effect on HIV-1 cell reservoirs of the concomitant administration of intensive chemotherapy and the pharmacological blockade of CCR5 coreceptors: a pilot, open, randomized, and controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give written consent to participate in the study
* Age between 18 and 65 years old, included.
* Chronic HIV-1 Demonstration of R5 viral tropism (use of CCR5 coreceptors) by genotyping in plasma samples stored
* Patients that are to be treated with intensive chemotherapy for non Hodgkin lymphoma With or without stable antiretroviral therapy
* Patients that are able to understand the purpose of the study and be available for scheduled appointments.
* Both in the case of female and male patients, the patient agrees to use a double barrier method of contraception from the moment of signing the informed consent until 3 months after the end of their participation in the study.

Exclusion Criteria:

* To have planned antiretroviral treatment interruption during the participation in the study
* Hypersensitivity to products used in this study
* To be involved in another clinical trial or received an investigational drug within 3 months prior to the study initiation
* To have contraindications or limitations to perform leukapheresis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
number of resting memory CD4+ T cells latently infected with replicative HIV-1, expressed as IUPM | Same as chemotherapy treatment (expected average of 6 months)
  Primary outcome will be measured before, during and after chemotherapy treatment until patient has reached normal lymphocytes levels

SECONDARY OUTCOMES:
Proviral DNA (copies/million cells) | Same as chemotherapy treatment (expected average of 6 months)
  Secondary outcome will be measured before, during and after chemotherapy treatment until patient has reached normal lymphocytes levels
Effector T cells producing HIV-1 specific gamma interferon (cells/mm3) | Same as chemotherapy treatment (expected average of 6 months)
  Secondary outcome will be measured before, during and after chemotherapy treatment until patient has reached normal lymphocytes levels
Levels of HIV-1 antibodies | Same as chemotherapy treatment (expected average of 6 months)
  Secondary outcome will be measured before, during and after chemotherapy treatment until patient has reached normal lymphocytes levels
Percentage of CD4+ and CD8+ cells with immune activation markers | Same as chemotherapy treatment (expected average of 6 months)
  Secondary outcome will be measured before, during and after chemotherapy treatment until patient has reached normal lymphocytes levels

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Ramon Y Cajal, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid

REFERENCES:
- [Background] Wang C, Vlahov D, Galai N, Bareta J, Strathdee SA, Nelson KE, Sterling TR. Mortality in HIV-seropositive versus -seronegative persons in the era of highly active antiretroviral therapy: implications for when to initiate therapy. J Infect Dis. 2004 Sep 15;190(6):1046-54. doi: 10.1086/422848. Epub 2004 Aug 17. PMID 15319852
- [Background] Moreno S, Mocroft A, Monforte Ad. Medical and societal consequences of late presentation. Antivir Ther. 2010;15 Suppl 1:9-15. doi: 10.3851/IMP1523. PMID 20442456
- [Background] Chun TW, Stuyver L, Mizell SB, Ehler LA, Mican JA, Baseler M, Lloyd AL, Nowak MA, Fauci AS. Presence of an inducible HIV-1 latent reservoir during highly active antiretroviral therapy. Proc Natl Acad Sci U S A. 1997 Nov 25;94(24):13193-7. doi: 10.1073/pnas.94.24.13193. PMID 9371822
- [Background] Finzi D, Hermankova M, Pierson T, Carruth LM, Buck C, Chaisson RE, Quinn TC, Chadwick K, Margolick J, Brookmeyer R, Gallant J, Markowitz M, Ho DD, Richman DD, Siliciano RF. Identification of a reservoir for HIV-1 in patients on highly active antiretroviral therapy. Science. 1997 Nov 14;278(5341):1295-300. doi: 10.1126/science.278.5341.1295. PMID 9360927